CLINICAL TRIAL: NCT01070888
Title: A Randomized, Double-blind, Double Dummy Crossover Trial on the Effect of Budesonide/Formoterol and Inhaled Budesonide Alone on Exercise-Induced Asthma in Patients With Persistent Asthma
Brief Title: Trial on the Effect of Budesonide/Formoterol and Inhaled Budesonide Alone on Exercise-Induced Asthma
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to reach target goal
Sponsor: Boston Children's Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Wanda Phipatanakul, Study PI, Boston Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08080372
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Results first posted 2014-12-30 (Estimated); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Exercise Induced Asthma
Keywords: Asthma; Exercise Induced Asthma
MeSH Terms: conditions — Asthma, Exercise-Induced; Asthma | interventions — Budesonide, Formoterol Fumarate Drug Combination; Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Budesonide/Formoterol first (Experimental): This arm will receive blinded budesonide/formoterol and dummy inhaler and will be asked to take 2 inhalations of each inhaler, twice daily. The second study period will be budesonide and dummy inhaler.
  Interventions: Drug: Budesonide/Formoterol; Drug: Budesonide
- Budesonide first (Active Comparator): This arm will receive blinded budesonide and dummy inhaler and will be asked to take 2 inhalations of each inhaler, twice daily. The second study period will be budesonide/formoterol and dummy inhaler.
  Interventions: Drug: Budesonide/Formoterol; Drug: Budesonide

INTERVENTIONS:
Drug: Budesonide/Formoterol — Budesonide/Formoterol 160/4.5, 2 puff twice daily for 2 weeks
  Other Names: Symbicort
Drug: Budesonide — Budesonide 180mcg, 2 puffs twice daily for 2 weeks
  Other Names: Pulmicort

SUMMARY:
The purpose of this study is to find out if Symbicort® (budesonide/formoterol), a new combination asthma medication, is more effective than budesonide alone in controlling exercise induced asthma.

The investigators hypothesize that in children and adults who suffer from asthma and exercise induced asthma there will be less decline in lung function associated with exercise when they receive the study medication.

DETAILED DESCRIPTION:
The purpose of this study is to find out if Symbicort® (budesonide/formoterol), a new combination asthma medication, is more effective than budesonide alone in controlling exercise induced asthma.

The investigators hypothesize that in children and adults who suffer from asthma and exercise induced asthma there will be less decline in lung function associated with exercise when they receive the study medication.

40 subjects will be randomized to receive both active medications in separate testing periods to determine the effect on their lung function after exercise testing.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female Patients aged 12 to 50 years with a diagnosis of asthma for at least 6 months before screening
* Baseline FEV1 of 60% to >100% of predicted
* Demonstrate a decrease in FEV1 of 15% or greater from baseline after standardized stepped exercise challenge testing
* Taking a constant dose of low-medium dose inhaled steroids for at least 30 days before screening of either:

  1. fluticasone, 88 - 440 mcg/d via MDI or 100 to 500 mcg/d via DPI
  2. beclomethasone HFA 80 to 480 mcg/day
  3. budesonide DPI 180 to 1200 mcg/ d
  4. flunisolide 500 to 2000 mcg/d
  5. flunisolide HFA 320 to 640 mcg/d
  6. mometasone 200 to 800 mcg/d
  7. triamcinolone acetonide 300 to 1500 mcg/ d

Exclusion Criteria:

* Patients already on LABAs, systemic corticosteroids, or other combination inhaled steroids/LABA medications.
* Patients not able to safely complete an exercise challenge due to physical constraints outside of their respiratory status.
* Patients who are pregnant or plan to become pregnant during the study period.
* Patients with a history of hypersensitivity reaction to either formoterol or budesonide.
* Patients with any significant disease or disorder which, in the opinion of the investigator, may either put the patient at risk because of participation in the study, or influence the results of the study, or the patient's ability to participate in the study.
* Patients with planned hospitalization during the study
* Current Smokers or those with a history of 10 pack years of tobacco use or more.

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2010-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wanda Phipatanakul, MD,MS, Principal Investigator — Boston Children's Hospital; Jonathan M Gaffin, MD, Study Director — Boston Children's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts

REFERENCES:
- [Derived] Gaffin JM, Bouzaher A, McCown M, Larabee Tuttle K, Israel E, Phipatanakul W. Rethinking the prevalence of exercise-induced bronchoconstriction in patients with asthma. Ann Allergy Asthma Immunol. 2013 Dec;111(6):567-8. doi: 10.1016/j.anai.2013.10.005. Epub 2013 Oct 30. No abstract available. PMID 24267370

RESULTS

PARTICIPANT FLOW:
Recruitment Details: October 2010 to October 2012
Pre-assignment Details: excluded from failed run-in or not qualify by exercise challenge
Groups:
- Budesonide First: This arm will receive blinded budesonide and dummy inhaler and will be asked to take 2 inhalations of each inhaler, twice daily. Subjects will subsequently take blinded budesonide/formoterol and dummy inhale, 2 inhalations of each, twice daily.
  Budesonide : Budesonide 180mcg, 2 puffs twice daily for 2 weeks
- Budesonide/Formoterol First: This arm will receive blinded budesonide/formoterol and dummy inhaler and will be asked to take 2 inhalations of each inhaler, twice daily. Subjects will subsequently take blinded budesonide and dummy inhale, 2 inhalations of each, twice daily.
  Budesonide/Formoterol : Budesonide/Formoterol 160/4.5, 2 puff twice daily for 2 weeks
Period: First Intervention (14 Days)
Arm/Group | Budesonide First | Budesonide/Formoterol First
Started | 2 | 4
Completed | 2 | 2
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Washout (14 Days)
Arm/Group | Budesonide First | Budesonide/Formoterol First
Started | 2 | 2
Completed | 1 | 2
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0
Period: Second Intervention (14 Days)
Arm/Group | Budesonide First | Budesonide/Formoterol First
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Budesonide First: This arm will receive blinded budesonide and dummy inhaler and will be asked to take 2 inhalations of each inhaler, twice daily.
  Budesonide first: Budesonide 180mcg, 2 puffs twice daily for 2 weeks, followed by a washout, then Budesonide/Formoterol 160/4.5, 2 puff twice daily for 2 weeks
- Budesonide/Formoterol First: This arm will receive blinded budesonide/formoterol and dummy inhaler and will be asked to take 2 inhalations of each inhaler, twice daily.
  Budesonide/Formoterol : Budesonide/Formoterol 160/4.5, 2 puff twice daily for 2 weeks, followed by a washout, then Budesonide 180mcg, 2 puffs twice daily for 2 weeks,
- Total: Total of all reporting groups
Arm/Group | Budesonide First | Budesonide/Formoterol First | Total
Number analyzed (Participants) | 2 | 4 | 6
Age, Continuous [Mean (Full Range); unit: years] | 29.5 [18 to 41] | 22.5 [15 to 33] | 24.8 [15 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 0 | 2 | 2
FEV1 fall % predicted with exercise [Mean (Standard Deviation); unit: percent fall in FEV1] | 15.5 (0.6) | 61.1 (13.0) | 45.9 (25.6)

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference Between Maximal Percentage Decrease in FEV1 After the Exercise Challenge Compared to the Run in Period, Budesonide/Formoterol - Budesonide
Description: Mean difference between maximal percentage decrease in FEV1 after the exercise challenge compared to the run in period, budesonide/formoterol - budesonide, calculated as follows:
  (max fall in FEV1(baseline) - maximal fall in FEV1(bud/form) - (max fall in FEV1(baseline) - maximal fall in FEV1(bud))
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: percentage of fall in FEV1
Groups:
- Budesonide First: This arm will receive blinded budesonide and dummy inhaler and will be asked to take 2 inhalations of each inhaler, twice daily. Then in the subsequent study period take budesonide/formoterol plus dummy inhaler 2 inhalations of each inhaler, twice daily
  Budesonide : Budesonide 180mcg, 2 puffs twice daily for 2 weeks
- Budesonide/Formoterol First: This arm will receive blinded budesonide/formoterol and dummy inhaler and will be asked to take 2 inhalations of each inhaler, twice daily, then in the subsequent period take budesonide and dummy inhaler 2 puffs twice daily.
  Budesonide/Formoterol : Budesonide/Formoterol 160/4.5, 2 puff twice daily for 2 weeks
Arm/Group | Budesonide First | Budesonide/Formoterol First
Number analyzed (Participants) | 1 | 2
percentage of fall in FEV1 | -3.1 (0) | -19.4 (30.5)

ADVERSE EVENTS:
Time Frame: Throughout entire study, 2 years
Groups:
- Budesonide/Formoterol: This arm will receive blinded budesonide/formoterol and dummy inhaler and will be asked to take 2 inhalations of each inhaler, twice daily.
  Budesonide/Formoterol: Budesonide/Formoterol 160/4.5, 2 puff twice daily for 2 weeks, followed by a washout, then Budesonide 180mcg, 2 puffs twice daily for 2 weeks
- Budesonide: This arm will receive blinded budesonide and dummy inhaler and will be asked to take 2 inhalations of each inhaler, twice daily.
  Budesonide: Budesonide 180mcg, 2 puffs twice daily for 2 weeks, followed by a washout, then Budesonide/formoterol 180mcg, 2 puffs twice daily for 2 weeks
Arm/Group | Budesonide/Formoterol | Budesonide
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 1/5 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Budesonide/Formoterol (N=5) | Budesonide (N=4)
asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — one subject had an asthma exacerbation requiring ED evaluation during the budesonide formoterol intervention. The subject recovered completely.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No